CLINICAL TRIAL: NCT03446261
Title: A Randomized, Multicenter, Open, Parallel, Phase 4 Study to Compare the Efficacy and Safety of Rosuvastatin/Ezetimibe Combination Therapy vs Rosuvastatin Monotherapy in Korean Patients With Type 2 Diabetes Mellitus and Hypercholesterolemia
Brief Title: Rosuvastatin/Ezetimibe vs Rosuvastatin in Korean Patients With Type 2 Diabetes Mellitus and Hypercholesterolemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC029
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes Mellitus; Hypercholesterolemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvamibe® Tab (Experimental): Rosuvamibe® Tab (rosuvastatin 5mg/ezetimibe 10mg) qd for 8 weeks
  Interventions: Drug: Rosuvamibe® Tab
- Monorova® Tab (Active Comparator): Monorova® Tab (rosuvastatin 10mg) qd for 8 weeks
  Interventions: Drug: Monorova® Tab

INTERVENTIONS:
Drug: Rosuvamibe® Tab — Rosuvastatin 5mg/ezetimibe 10mg qd for 8 weeks
  Arms: Rosuvamibe® Tab
Drug: Monorova® Tab — Rosuvastatin 10mg qd for 8 weeks
  Arms: Monorova® Tab

SUMMARY:
To assess the efficacy and safety of rosuvastatin/ezetimibe combination therapy compared to rosuvastatin monotherapy in Korean patients with type 2 diabetes mellitus and hypercholesterolemia

DETAILED DESCRIPTION:
This study is to assess the efficacy and safety of Rosuvamibe® (rosuvastatin 5mg/ezetimibe 10mg) vs Monorova® (rosuvastatin 10mg) treated for 8 weeks in Korean patients with type 2 diabetes mellitus and hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19 to 70 years
2. Patient with type 2 diabetes who needs treatment for hypercholesterolemia
3. Written informed consent

Exclusion Criteria:

1. Administration of lipid lowering agents for more than one week within 4 weeks prior to screening visit
2. Uncontrollable diabetes with HbA1c ≥ 8.5%
3. Fasting LDL-C ≤ 70 mg/dL
4. Fasting triglyceride ≥ 400 mg/dL
5. Total cholesterol ≥ 300 mg/dL
6. History of muscular disease or rhabdomyolysis due to use of statin
7. Hypersensitive to rosuvastatin or ezetemibe
8. Contraindications stated in the SPC of rosuvastatin or rosuvastatin/ezetimibe including the following:

   ① Severe renal disease (estimated GFR(MDRD) < 30mL/min/1.73m2)

   ② ALT, AST > 3x ULN or history of active liver disease

   ③ CPK > 3x ULN
9. Administration of other investigational products within 30 days prior to screening visit
10. Other than the above who is deemed to be ineligible to participate in the trial by investigator

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 8 in ApoB/ApoA1 ratio | Baseline, Week 8

SECONDARY OUTCOMES:
Proportion of over 50% reduction in LDL-C | Baseline, Week 8
Proportion of subjects achieving the comprehensive lipid target (LDL-C<70mg/dL, Non-HDL-C<100mg/dL, and ApoB<80mg/dL) | Baseline, Week 8
Change from baseline to week 8 in total, non-HDL, LDL and HDL cholesterol, triglyceride, ApoB, ApoA1 and ApoB48 | Baseline, Week 8
Change from baseline to week 8 in HOMA-IR | Baseline, Week 8
Change from baseline to week 8 in hs-CRP | Baseline, Week 8
Change from baseline to week 8 in HbA1C | Baseline, Week 8
Change from baseline to week 8 in FPG | Baseline, Week 8

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Asan Medical Center, Kora-ri
  - Asan Medical Center, Seoul

REFERENCES:
- [Derived] Lee J, Hwang YC, Lee WJ, Won JC, Song KH, Park CY, Ahn KJ, Park JY. Comparison of the Efficacy and Safety of Rosuvastatin/Ezetimibe Combination Therapy and Rosuvastatin Monotherapy on Lipoprotein in Patients With Type 2 Diabetes: Multicenter Randomized Controlled Study. Diabetes Ther. 2020 Apr;11(4):859-871. doi: 10.1007/s13300-020-00778-1. Epub 2020 Feb 17. PMID 32065359